CLINICAL TRIAL: NCT05300061
Title: Evaluating the Use of Brief Values Interventions in Increasing Willingness to Approach and Approach Behaviour Towards Phobic Stimuli in Specific Phobias
Brief Title: Values Interventions for Increasing Engagement With What is Feared in Individuals With Specific Phobias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Collaborators: Youth Board of Cyprus (Unknown)
Responsible Party: Principal Investigator, Maria Karekla, Associate Professor, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K3_K1_3
Record Dates: First submitted 2021-11-24; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Specific Phobia
Keywords: Specific Phobia; Flying Phobia; Exposure Therapy; Values Interventions
MeSH Terms: conditions — Phobia, Specific; Aerophobia

STUDY DESIGN:
Intervention Model Description: Three-arm randomised control trial including two values interventions: (a) a personal one, b) a prosocial one, and (c) a no-instructions control. Each participant is allocated to one of the three arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personal Values Intervention (Experimental): Brief personal values intervention
  Interventions: Behavioral: Personal Values Intervention
- Prosocial Values Intervention (Experimental): Brief prosocial values intervention
  Interventions: Behavioral: Prosocial Values Intervention
- Control (No Intervention): No intervention control

INTERVENTIONS:
Behavioral: Personal Values Intervention — A 15 minute personal values intervention. Aim is to help participants clarify their own values around flying and promote committed action towards airplanes.
  Arms: Personal Values Intervention
Behavioral: Prosocial Values Intervention — A 15 minute prosocial values intervention. Aim is to help participants clarify their prosocial values around flying and promote committed action towards airplanes.
  Arms: Prosocial Values Intervention

SUMMARY:
Exposure is considered the therapy of choice for specific phobias (SPs). Nevertheless, therapy engagement is extremely limited. SPs are maintained through avoidance of feared stimuli and as such willingness to approach what is feared constitutes a key factor that could explain limited treatment engagement. Values interventions, a key element of acceptance and commitment therapy (ACT), might be one way to increase engagement, yet to this date limited research exists in this area. For the purposes of the current study, two brief values interventions were developed: (a) a personal and (b) a prosocial one. These will be compared to (c) a no-instructions control in increasing willingness to approach and approach behaviour towards phobic stimuli. Ninety participants with flying phobia will be randomly allocated to one of the three groups. To measure willingness to engage with feared stimuli and approach behaviour two behavioural approach tasks using novel technologies (virtual reality), which aimed to expose participants to situations analogous to real life, were developed. Willingness and behavioural approach towards airplanes at a one month follow up will also be assessed.

Therefore, it is hypothesised that:

1. Participants in either of the two values intervention groups will have greater willingness to engage and approach behaviour towards feared stimuli compared to those in control, during the study tasks.
2. Participants in either of the two values intervention groups will have greater willingness to engage and approach behaviour towards feared stimuli compared to those in control at follow up.

   Additionally, as prosocial values provide an evolutionary advantage, the second study aim was to identify if they lead to greater engagement with phobic stimuli compared to personal ones. Therefore, it was also hypothesised that:
3. Participants in the prosocial values group will have greater willingness to engage and approach behaviour towards feared stimuli compared to those in personal values group, both during the study tasks and at follow up.
4. Participants in the prosocial values group will have greater willingness to engage and approach behaviour towards feared stimuli compared to those in personal values group at follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Meeting the Diagnostic and Statistical Manual for Mental Disorders 5
* Good knowledge of the Greek language (adequate comprehension level, reading level, and verbal communication)

Exclusion Criteria:

* Severe heart disease
* High blood pressure
* Photosensitive epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Willingness | Day 1 (During experimental tasks)
  In order to capture willingness to engage with feared stimuli three questions were employed, one question for each study task and one for follow up. For example to capture willingness to engage with the virtual reality behavioural approach task, participants were asked: "How willing are you to participate in a virtual reality task involving airplanes?". Answers for all three questions were rated on a scale from 1 (Not willing at all) to 10 (Extremely willing), with higher scores indicating greater willingness levels (i.e., total score: 1 - 10). This approach for developing willingness questions was based on other studies similarly aiming to capture willingness as part of their outcomes using a brief measure (e.g., Fink-Lamotte et al., 2020).
Virtual Reality Behavioural Approach Task (VR BAT) | Day 1 (During experimental tasks)
  The virtual reality (VR) behavioural approach task was developed for the current study to capture approach behaviour towards airplanes in VR. In total the task included seven steps. Each step depicted a different aspect of flying with associated VR visuals and sounds: 1) airplane stopped engine off, 2) airplane stopped engine running, 3) taxiing, 4) take off, 5) cruising, 6) turbulence and 7) landing, each lasting between 51 and 129 seconds. Approach behaviour was calculated by adding the number of steps participants completed in the VR BAT with total approach behaviour score ranging from 0 to 7.
Behavioural Willingness Assessment (BWA) | Day 1 (During experimental tasks)
  For this task, participants were presented with the option to book a short complementary flight. This was a categorical response variable: Participants could either book a flight or decline to participate. Booking a flight indicated approach behaviour towards airplanes.
Follow up Flying Behaviour | One month follow up
  To measure approach behaviour towards airplanes outside the laboratory setting at a one month follow up, one question was employed ("In the past month, have you come in contact with airplanes in any way, such as taking a flight, or booking flight tickets or hotels abroad?") with a "yes" or "no" response (categorical response variable). An affirmative response indicated approach behaviour towards airplanes.

SECONDARY OUTCOMES:
Avoidance Behaviours | Day 1 (During experimental tasks)
  Total number of avoidance behaviours employed by the participants during the virtual reality behavioural approach task were tallied by the experimenter.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Karekla, PhD, Principal Investigator — University of Cyprus
Locations (1):
- University of Cyprus, Nicosia, Non-US/Non-Canadian, Cyprus

IPD SHARING:
Plan to Share IPD: No